CLINICAL TRIAL: NCT06485752
Title: A Phase 3, Randomized, Observer-Blinded, Study to Compare the Safety and Immunogenicity of 3 Lots of Trivalent Hemagglutinin Nanoparticle Influenza Vaccine With Matrix M™ Adjuvant in Participants ≥ 60 Years of Age
Brief Title: Phase 3 Lot Consistency Study of Trivalent Hemagglutinin Nanoparticle Influenza Vaccine
Status: Withdrawn | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: Decided to not move forward with the study
Sponsor: Novavax (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Prevention
Other Study IDs: tNIV-E-316
Record Dates: First submitted 2024-06-27; First posted 2024-07-03 (Actual); Last update posted 2025-03-11 (Actual); Status verified 2025-03

CONDITIONS: COVID-19
Keywords: COVID-19, influenza Vaccine
MeSH Terms: conditions — COVID-19; Influenza, Human | interventions — Influenza Vaccines

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Lot 1 (Group 1) (Active Comparator): influenza A [H1N1]
  Interventions: Biological: tNIV 1 and Matrix-M Adjuvant
- Lot 2 (Group 2) (Active Comparator): influenza A [H3N2]
  Interventions: Biological: tNIV 1 and Matrix-M Adjuvant
- Lot 3 (Group 3) (Active Comparator): influenza B-Victoria lineage strains
  Interventions: Biological: tNIV 1 and Matrix-M Adjuvant

INTERVENTIONS:
Biological: tNIV 1 and Matrix-M Adjuvant — tNIV will be administered as a single 0.5 mL IM injection Day 0
  Other Names: Influenza vaccine

SUMMARY:
Phase 3 Study Comparing Safety and Immune Response of Three Batches of Novavax Flu Vaccine in older adult participants

DETAILED DESCRIPTION:
This is a randomized, Phase 3 study comparing the safety and immunogenicity of 3 different lots of Novavax trivalent hemagglutinin (HA) nanoparticle influenza vaccine (NIV) with Matrix-M (tNIV) in terms of wild-type influenza hemagglutinin inhibition (HAI) antibody responses to 3 vaccine-homologous influenza strains (ie, 2 influenza A strains and an influenza B-Victoria lineage strain).

ELIGIBILITY:
Inclusion Criteria:

* To be included in this study, each individual must satisfy all of the following criteria:

  1. Willing and able to give informed consent prior to study enrollment.
  2. Medically stable adult male or female ≥ 60 years of age at Screening.
  3. Participants may have 1 or more chronic medical diagnoses, but should be clinically stable as assessed by:

     1. Absence of changes in medical therapy in the past 2 months due to treatment failure or toxicity;
     2. Absence of medical events qualifying as SAEs within 3 months; and
     3. Absence of known, current, and life-limiting diagnoses which render survival to completion of the protocol unlikely in the opinion of the Investigator.
  4. The participant has a body mass index (BMI) of 17 to 40 kg/m2, inclusive, at Screening.
  5. Participant must be able to receive an injection in the deltoid of at least one arm.
  6. Able to attend study visits, comply with study requirements, and provide reliable and complete reports of AEs.
  7. Women of childbearing potential (defined as any female participant who is NOT surgically sterile [ie, hysterectomy, bilateral tubal ligation, or bilateral oophorectomy] or postmenopausal [defined as amenorrhea at least 12 consecutive months]) must agree to be heterosexually inactive from at least 28 days prior to enrollment and through the end of the study OR agree to consistently use a medically acceptable method of contraception listed below from at least 28 days prior to enrollment and through the end of the study.

     1. Condoms (male or female) with spermicide (if acceptable in country)
     2. Diaphragm with spermicide
     3. Cervical cap with spermicide
     4. Intrauterine device
     5. Oral or patch contraceptives
     6. Norplant®, Depo-Provera®, or other in-country regulatory approved contraceptive method that is designed to protect against pregnancy
     7. Abstinence as a form of contraception, is acceptable if in line with the participant's lifestyle
  8. Participants must agree to not participate in any other severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2) or influenza prevention or treatment studies for the duration of the study. Note: For participants who become hospitalized with COVID-19 or influenza, participation in investigational treatment studies is permitted.

Exclusion Criteria:

* If an individual meets any of the following criteria, he or she is ineligible for this study:

  1. Any ongoing, symptomatic acute illness requiring medical or surgical care or chronic illness that required substantive changes in medication in the past 2 months prior to Screening indicating that chronic illness/disease is not stable (at the discretion of the Investigator). This includes any current workup of undiagnosed illness that could lead to a new condition.
  2. Serious chronic diseases inclusive of:

     1. Uncontrolled hypertension (NOTE: hypertension ≤ 170/100 is NOT exclusionary);
     2. Congestive heart failure requiring hospitalization within 3 months prior to Screening (NOTE: stable congestive heart failure is NOT exclusionary);
     3. Chronic obstructive pulmonary disease (COPD) requiring hospitalization within 3 months prior to Screening (NOTE: stable COPD is NOT exclusionary);
     4. Within 3 months prior to Screening, evidence of unstable coronary artery disease as manifested by cardiac interventions (eg, cardiac stent placement, coronary artery bypass graft surgery), new cardiac medications for control of symptoms, or unstable angina (NOTE: stable coronary heart disease is NOT exclusionary);
     5. Hospitalization for diabetic ketoacidosis within 6 months prior to Screening
     6. Chronic kidney disease/renal requiring institution of substantive new therapy within 3 months prior to Screening
     7. Chronic clinically significant gastrointestinal and hepatic diseases requiring hospitalization or institution of substantive new therapy within 3 months prior to Screening. (f or example, gastroesophageal reflux disease is NOT exclusionary)
     8. Chronic neurological diseases or neurological compromise preventing access to the study clinic, compliance with protocol, or accurate reporting of safety.
  3. Participation in research involving an investigational product (drug/biologic/device) within 90 days before planned date of vaccination.
  4. Use of COVID-19 prophylactic or treatment monoclonal antibodies or antibody cocktails within 90 days prior to planned date of vaccination.
  5. History of a serious reaction to a prior influenza vaccination or known allergy to constituents of influenza vaccines - including egg proteins - or polysorbate 80; or any known allergies to products contained in the investigational product.
  6. Any history of anaphylaxis to any prior vaccine.
  7. History of Guillain-Barré Syndrome within 6 weeks following a previous influenza vaccine.
  8. Receipt of any vaccine in the 4 weeks preceding the study vaccination and any influenza vaccine within 2 months preceding the study vaccination. Note: Routine vaccinations will not be allowed until after study Day 28 and COVID-19 and influenza vaccination will not be allowed until after Day 28.
  9. Any known or suspected autoimmune or immunosuppressive illness, congenital or acquired, based on medical history and/or physical examination (NOTE: well-controlled hypothyroidism and mild psoriasis are not exclusionary).
  10. Chronic administration (defined as more than 14 continuous days) of immunosuppressants or other immune-modifying drugs within 6 months prior to the administration of the study vaccines. An immunosuppressant dose of glucocorticoid is defined as a systemic dose ≥ 10 mg of prednisone per day or equivalent. The use of topical, inhaled, and nasal glucocorticoids is permitted.
  11. Administration of immunoglobulins and/or any blood products within the 3 months preceding the administration of the study vaccine or during the study.
  12. Active cancer (malignancy) therapy within 1 year prior to study vaccination (with the exception of adequately treated non-melanomatous skin carcinoma or lentigo maligna and uterine cervical carcinoma in situ without evidence of disease, at the discretion of the Investigator).
  13. Participants who are breastfeeding, pregnant, or who plan to become pregnant prior to the EoS.
  14. Suspected or known history of alcohol abuse or drug addiction within 2 years prior to study vaccination, which in the opinion of the Investigator, might interfere with protocol compliance.
  15. Acute disease at the time of enrollment (defined as the presence of a moderate or severe illness with or without fever, or an oral temperature ≥ 38.0°C, on the planned day of vaccine administration).
  16. Any condition that in the opinion of the Investigator would pose a health risk to the participant if enrolled or could interfere with evaluation of the vaccine or interpretation of study results (including neurologic or psychiatric conditions deemed likely to impair the quality of safety reporting).
  17. Study team member or immediate family member of any study team member (inclusive of Sponsor, contract research organization, and study site personnel involved in the conduct or planning of the study).

Ages: 60 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2024-11 (Estimated); Primary Completion 2025-02-04 (Actual); Study Completion 2025-02-04 (Actual)

PRIMARY OUTCOMES:
Safety- Solicited AEs over 7 days post-vaccination | 7 days post-vaccination
  Numbers and proportions of participants with solicited local and systemic AEs over the 7 days post-vaccination.
Safety- Unsolicited AEs and MAAEs over 28 days post-vaccination | Day 0 to 28
  Numbers and proportions of participants reporting unsolicited AEs and MAAEs over 28 days post-vaccination.
Safety-Treatment-related MAAEs, SAEs, and AESIs (including PIMMC) | Day-0 to 182
  Numbers and proportions of participants with treatment-related MAAEs, AESIs (including PIMMCs), and SAEs over 6 months (approximately 182 days) post-vaccination.
Immunogenicity-HAI antibody titers specific for the HA receptor binding domains of vaccine homologous A and B influenza strains Expressed as GMT | Day-0 to 28
  HAI antibody titers specific for the HA receptor binding domains of vaccine response to 3 vaccine-homologous influenza strains (ie, 2 influenza A strains and an influenza B-Victoria lineage strain) at Day 28.
Immunogenicity-HAI antibody titers specific for the HA receptor binding domains of vaccine homologous A and B influenza strains Expressed as GMTR | Day-0 to 28
  HAI antibody titers specific for the HA receptor binding domains of vaccine response to 3 vaccine-homologous influenza strains (ie, 2 influenza A strains and an influenza B-Victoria lineage strain) at Day 28.

SECONDARY OUTCOMES:
Influenza NAb responses: neutralizing antibody titers specific to vaccine homologous wild-type A and B influenza strains, is expressed as GMT | Day 0 to Day 28
  Neutralizing antibody titers specific to vaccine homologous wild-type A and B influenza strains, as measured by a neutralization assay of vaccine response to 3 vaccine-homologous influenza strains (ie, 2 influenza A strains and an influenza B-Victoria lineage strain) at Day 28.
Influenza NAb responses: neutralizing antibody titers specific to vaccine homologous wild-type A and B influenza strains, is expressed as GMTR | Day 28 [Post vaccination]
  Neutralizing antibody titers specific to vaccine homologous wild-type A and B influenza strains, as measured by a neutralization assay of vaccine response to 3 vaccine-homologous influenza strains (ie, 2 influenza A strains and an influenza B-Victoria lineage strain) at Day 28 [Post vaccination].
Influenza NAb responses: neutralizing antibody titers specific to vaccine homologous wild-type A and B influenza strains, is expressed as SCR | Day 28 [Post vaccination]
  Neutralizing antibody titers specific to vaccine homologous wild-type A and B influenza strains, as measured by a neutralization assay of vaccine response to 3 vaccine-homologous influenza strains (ie, 2 influenza A strains and an influenza B-Victoria lineage strain) at Day 28 [Post vaccination].